CLINICAL TRIAL: NCT06722885
Title: Observational Study of Stereotactic Body Radiotherapy for Lung Lesions With Markerless Tracking (MLT) on the VERO® SBRT System
Brief Title: Stereotactic Body Radiotherapy for Lung Lesions With Markerless Tracking (MLT) on the VERO® SBRT System
Acronym: SBRT_LOV
Status: Withdrawn | Type: Observational
Why Stopped: The VERO® SBRT System radiation machine had water damage and could not be repaired.
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Mark De Ridder, Prof Dr, Universitair Ziekenhuis Brussel
Other Study IDs: SBRT_LOV
Record Dates: First submitted 2019-05-14; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Stereotactic Body Radiotherapy; Lung Diseases; Lung Cancer Metastatic; Lung Cancer Stage IV; Lung Cancer, Nonsmall Cell
Keywords: radiotherapy; stereotactic body radiotherapy; markerless tracking; clinical feasibility; implementation
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Markerless tracking: * Gross tumor volume for MLT (GTV_MLT): lesion delineated on stable exhale phase of the 4DCT.
  * Planning target volume for MLT (PTV_MLT): GTV + 8 mm isotropic expansion
  Interventions: Radiation: Standard radiotherapy treatment
- ITV approach: * Gross tumor volume (GTV): lesion delineated on the ten phases of the 4DCT.
  * Internal target volume (ITV): propagate all GTV on stable exhale phase of the 4DCT.
  * Planning target volume for ITV (PTV_ITV): ITV + 5 mm isotropic expansion
  Interventions: Radiation: Standard radiotherapy treatment
- Markerbased tracking: * Gross tumor volume for tracking (GTV_Track): lesion delineated on stable exhale phase of the 4DCT.
  * Planning target volume for tracking (PTV_Track): GTV + 5 mm isotropic expansion
  Interventions: Radiation: Standard radiotherapy treatment

INTERVENTIONS:
Radiation: Standard radiotherapy treatment — * 3 x 17 Gy for peripheral NSCLC
  * 4 x 12 Gy in centrally located NSCLC or at < 1cm from the thoracic wall
  * 8 x 7,5 Gy if with the predefined dose for NSCLC, the constraints of the organs at risk cannot be met
  * 5 x 8,5 Gy in case of oligometastases

SUMMARY:
Stereotactic Body Radiotherapy (SBRT) delivers an ablative dose of radiation to tumours, with high precision. This technique offers an alternative to surgery for lung lesions. The UZ Brussel of the VUB developed with the support of the Hercules foundation (grant for heavy research infrastructure) in collaboration with Brainlab AG a breathing-synchronized radiation technique on the VERO SBRT system, where the radiation beam follows the moving target (dynamic tumour tracking). The implantation of a marker in the tumour is thereby mandatory for its visualization but excluding patients with poor pulmonary function. Therefore Brainlab® recently released an update of the VERO SBRT system that allows "Markerless Tracking". This markerless technique is currently being implemented at the Radiotherapy Department of UZ Brussel for lung lesions. Hence we plan an observational study that will document the outcome of and feasibility for patients with lung lesions treated with markerless tracking on the VERO SBRT system at the Radiotherapy Department in UZ Brussel.

DETAILED DESCRIPTION:
Stereotactic Body Radiotherapy (SBRT) delivers an ablative dose of radiation to tumours, with high precision. This technique offers an alternative to surgery for lung lesions. The movement of these tumours represents a clinical problem and a technological challenge. The UZ Brussel of the VUB developed with the support of the Hercules foundation (grant for heavy research infrastructure) in collaboration with Brainlab AG a breathing-synchronized radiation technique on the VERO SBRT system, where the radiation beam follows the moving target (dynamic tumour tracking). The implantation of a marker in the tumour is thereby mandatory for its visualization but excluding patients with poor pulmonary function. Moreover, the placement of such an implanted fiducial marker is contraindicated for about 30% of the patients and may be associated with complications such as pneumothorax and bleeding.

Therefore Brainlab® recently released an update of the VERO SBRT system that allows "Markerless Tracking" (MLT). This markerless technique is currently being implemented at the Radiotherapy Department of UZ Brussel for lung lesions. Within the Spearhead Strategic Research Program "Societal Benefit of Markerless Stereotactic Body Radiotherapy: a Statistical Support based on Quantitative Imaging", the investigators aim at evaluating the implementation of this technique focusing on patient outcomes and clinical feasibility. In order to do so they plan an observational study that will document the feasibility and outcome of patients with lung lesions treated with markerless tracking on the VERO SBRT system at the Radiotherapy Department in UZ Brussel.

ELIGIBILITY:
Inclusion Criteria:

1. Primary NSCLC patients, stage T1-2bN0M0 (TNM 8th edition)
2. Oligometastatic patients with ≤ 3 lung metastases; SBRT as a primary treatment or as a consolidative treatment after induction chemotherapy;
3. >= 18 years
4. Patients will be recruited via the treating radiotherapist

   -

   Exclusion Criteria:

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung lesions or primary lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of patients treated with markerless and markerbased technique | 1 week
  Comparing patient characteristics between markerbased and marker less technique
Local tumor control | 1 year
  local control at 1 year
Number of patients with acute toxicity | up to 6 months
  according to Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0)
Number of patients with late toxicity | up to 5 years
  according to Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0)
Disease free survival | up to 5 years
  Disease free survival
Overall survival | up to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Mark De Ridder, MD, PhD, Study Chair — Universitair Ziekenhuis Brussel; Christine Collen, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided